CLINICAL TRIAL: NCT01473056
Title: Phase I,Randomized,Double-blind,Placebo-controlled,Multiple Dose Study Evaluating Safety,Tolerability,Pharmacokinetics and Antiviral Activity of JTK-853 in HCV Genotype 1 Infected Subjects,Followed by a Genotypic Resistance Monitoring Study
Brief Title: Study to Assess Safety,Tolerability,Pharmacokinetics & Antiviral Activity of JTK-853 in Hepatitis C Virus Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK853-U-09-002
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of
Keywords: Hepatitis C; JTK-853
MeSH Terms: conditions — Hepatitis C | interventions — JTK-853

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose 1 JTK-853 (Experimental)
  Interventions: Drug: JTK-853
- Dose 2 JTK-853 (Experimental)
  Interventions: Drug: Dose 2 JTK-853
- Dose 3 JTK-853 (Experimental)
  Interventions: Drug: Dose 3 JTK-853
- Dose 4 JTK-853 (Experimental)
  Interventions: Drug: Dose 4 JTK-853
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTK-853 — Tablets, twice a day for 3 days
  Arms: Dose 1 JTK-853
Drug: Dose 2 JTK-853 — Tablets, twice a day for 3 days
  Arms: Dose 2 JTK-853
Drug: Dose 3 JTK-853 — Tablets, three times a day for 3 days
  Arms: Dose 3 JTK-853
Drug: Dose 4 JTK-853 — Tablets, twice a day for 3 days
  Arms: Dose 4 JTK-853
Drug: Placebo — Tablets, twice a day or three times a day for 3 days
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the safety, tolerability, pharmacokinetics and anti-viral activity of JTK-853 in hepatitis C virus genotype 1 infected subjects based on reduction in viral load (HCV RNA level) from baseline to end of treatment, followed by genotypic resistance monitoring for up to one year after study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females infected with chronic hepatitis C virus (HCV) infection and genotype 1a or 1b
2. Subjects with a viral load (HCV RNA level) of ≥50,000 IU/mL
3. Subjects with a body mass index (BMI) of 18.0-36.0 kg/m2 (inclusive)

Exclusion Criteria:

1. Subjects should not have previously received a direct acting anti-HCV agent
2. Subjects should not previously have received pegylated interferon/ribavirin for a duration of more than two weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 1 week
Maximum concentration (Cmax) of JTK-853 and metabolite M2 | 1 week
Time to reach maximum concentration (tmax) for JTK-853 and metabolite M2 | 1 week
Area under the concentration-time curve during the dosing interval (AUCtau) for JTK-853 and Metabolite M2 | 1 week
Trough concentration during multiple dosing prior to next dose (Ctrough) for JTK-853 and metabolite M2 | 1 week
Viral load change from baseline to end of treatment | 48 weeks
Genotypic resistance assessment and viral load change from baseline over time | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Hoshino, D.V.M, Study Director — Akros Pharma Inc.
Locations (1):
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico